CLINICAL TRIAL: NCT06186362
Title: Clinical and Radiological Results of Distal Clavicle Auto Graft in Patient With Recurrent Anterior Shoulder Dislocation
Brief Title: Results of Distal Clavicle Graft in Shoulder Dislocation Clavicle Auto Graft in Patient With Recurrent Anterior Shoulder Dislocation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mostafa Khalaf Mahmoud Mohammed, Principle investigator, Al-Azhar University
Other Study IDs: DCRSD
Record Dates: First submitted 2023-11-20; First posted 2024-01-02 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Shoulder Injuries
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
to evaluate the clinical and radiological Outcome of Distal Clavicle Auto graft in patient with recurrent Shoulder dislocation

DETAILED DESCRIPTION:
The glenohumeral joint is the most commonly dislocated joint of the human body,The stability of GH joint relies on a complex network of static and dynamic structures,The anterior labrum plays a key role in antero posterior stability as it deepens the glenoid cavity up to 50% There option for glenoid reconstruction including: Distal Clavicle Auto graft (DCA), proven is a good option to coracoid transfers

ELIGIBILITY:
Inclusion Criteria:

* Recurrent Traumatic anterior shoulder dislocation (≥ 3 times).

Exclusion Criteria:

.On-track Hill-Sachs lesion. .Multi directional instability.

* Voluntary dislocation.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Range of motion "ROM" (Forward flexion, external rotation, internal rotation) Preoperative and postoperative ROM . Rowe score, Visual analogue score (VAS). Secondary outcomes postoperative complications will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Row score | At 2 months, 6 months post operative
  Rang of motion

REFERENCES:
- [Background] Kane P, Bifano SM, Dodson CC, Freedman KB. Approach to the treatment of primary anterior shoulder dislocation: A review. Phys Sportsmed. 2015 Feb;43(1):54-64. doi: 10.1080/00913847.2015.1001713. Epub 2015 Jan 6. PMID 25559018